CLINICAL TRIAL: NCT01650454
Title: Sleep, Cognition and Memory Disorder
Acronym: SCOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2012/02
Record Dates: First submitted 2012-07-18; First posted 2012-07-26 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Sleep Architecture; Sleep Disorders; Cognitive Impairment
Keywords: Alzheimer; Sleep; Somnolence
MeSH Terms: conditions — Sleep Wake Disorders; Cognitive Dysfunction; Sleepiness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Patients from Memento cohort. (Experimental): Patients with mild cognitive impairment included in MEMENTO cohort.
  These patients will have a 2 night polysomnography, a battery of neuropsychological tests, a virtual reality test, and a subjective evaluation of sleep and somnolence at inclusion (Month 0) and Month 12.
  Interventions: Other: 2 night polysomnography; Other: battery of neuropsychological tests; Other: virtual reality test; Other: subjective evaluation of sleep and somnolence
- Patients with memory disorders (Experimental): Patients with mild cognitive impairment not included in MEMENTO cohort. For these patients a virtual reality test, and a subjective evaluation of sleep and somnolence will be performed at Inclusion (Month 0)
  Interventions: Other: virtual reality test; Other: subjective evaluation of sleep and somnolence
- Healthy volunteers (Active Comparator): Healthy volunteers matched in age, sex and educational level with patients. For these volunteers a virtual reality test, and a subjective evaluation of sleep and somnolence will be performed at Inclusion (Month 0)
  Interventions: Other: virtual reality test; Other: subjective evaluation of sleep and somnolence
- control group (Active Comparator): this group is composed with Healthy volunteers these volunteers will have a 2 night polysomnography, a battery of neuropsychological tests, a virtual reality test, and a subjective evaluation of sleep and somnolence at inclusion (Month 0) and Month 12.
  Interventions: Other: 2 night polysomnography; Other: battery of neuropsychological tests; Other: virtual reality test; Other: subjective evaluation of sleep and somnolence

INTERVENTIONS:
Other: 2 night polysomnography — Polysomnography
  Arms: Patients from Memento cohort.; control group
Other: battery of neuropsychological tests
  Arms: Patients from Memento cohort.; control group
Other: virtual reality test
Other: subjective evaluation of sleep and somnolence

SUMMARY:
The increasing incidence of Alzheimer's disease (AD) and related sleep-disorders with the aging of the population is a major issue of public health. The prevalence of sleep disturbances is about 50% in dementia patients. Sleep in dementia is mainly characterized by prolonged night-time awakenings, sometimes with longer sleep latency and/or early awakening. The presence of these sleep disturbances is the main reason for the institutionalization of AD patients, as well as a major cause of the deterioration of the caregivers' sleep. The MEMENTO cohort is composed of patients with isolated memory complaints or mild cognitive impairment, at high risk to develop dementia. All voluntary patients from the CMRR (Center of Memory, resources and Research) of Bordeaux (MEMENTO cohort) will be tested at inclusion and followed-up 1 year later. For these two evaluations, actigraphic monitoring at home, 2-night polysomnography (PSG) monitoring at hospital including a 24-hour period of urinary melatonin dosage, neuropsychological tests battery, a virtual reality tool and questionnaires will be used.

ELIGIBILITY:
Inclusion criteria for patients with mild cognitive impairment included in MEMENTO cohort:

* Aged 18 years and above
* included in MEMENTO cohort within the last 3 months
* Clinical dementia rating scale ≤ 0,5 (not demented)
* Patients with mild cognitive impairment
* Visual and auditory acuity adequate for neuropsychological testing
* Having signed an informed consent
* Being affiliated to health insurance

Inclusion criteria for patients with mild cognitive impairment not included in MEMENTO cohort:

* Aged 18 years and above
* First contact with Memory clinic within the last 3 months
* Clinical dementia rating scale ≤ 0,5 (not demented)
* Patients with mild cognitive impairment
* Visual and auditory acuity adequate for neuropsychological testing
* Having signed an informed consent
* Being affiliated to health insurance

Inclusion criteria for Healthy volunteers and Control group:

* Aged 18 years and above
* Without evidence of psychopathology
* Volunteers matched in age, sex and educational level with patients
* Visual and auditory acuity adequate for neuropsychological testing
* Having signed an informed consent
* Being affiliated to health insurance

Exclusion criteria:

* Being under guardian conservator
* Residence in skilled nursing facility
* Pregnant or breast feeding woman
* Alzheimer's disease caused by gene mutations
* Having a neurological disease
* History of stroke within the past three months
* Generalized anxiety (DSM-IV criteria)
* Schizophrenia history (DSM-IV criteria)
* Illiteracy, is unable to count or to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10-29 (Actual); Study Completion 2015-10-29 (Actual)

PRIMARY OUTCOMES:
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Apnea/Hypopnea index, periodic limb movements index
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Excessive transient muscle activity, Sustained muscle activity
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Sleep structure parameters (% stage 1, 2, 3 and Rapid Eye movement, Delta activity, Spindle rate)
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Sleep duration parameters
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Sleep consolidation parameters
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  - Sleep propensity parameters 24-hour melatonin quantity rate
Polysomnography of night 1 | Change from inclusion (Month 0) and Month 12
  Actimetry: Inter-daily stability, intra-daily variability, rhythm amplitude

SECONDARY OUTCOMES:
Subjective evaluation of sleep and Somnolence | Month 0 and Month 12
Evaluation of Memory disorder | Month 0 and Month12
  Reaction times and % of errors in the neuropsychological tests (memory, speed processing, language, visuo-spatial skills, attentional functions, executive functions)
Evaluation of Memory disorder | Month 0 and Month12
  % of recall from the memory test in a virtual environment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Philip, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France